CLINICAL TRIAL: NCT00475371
Title: A Phase 1a, Single-Dose, Open-Label, Parallel, Ascending Dose, Controlled Safety and Tolerability Trial of Inhaled MKC253 in Healthy Adult Male Subjects
Brief Title: A First in Human, Single Dose, Safety and Tolerability Study of MKC253 Inhalation Powder in Healthy Adult Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MKC-253-001; EudraCT Number 2007-000361-37
Record Dates: First submitted 2007-05-16; First posted 2007-05-21 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Diabetes Mellitus, Type 2; Healthy Males
Keywords: Healthy; Diabetes Mellitus: Type II
MeSH Terms: conditions — Diabetes Mellitus, Type 2

ARMS (1):
- 1 (Experimental): MKC253 Inhalation Powder
  Interventions: Drug: MKC253 Inhalation Powder

INTERVENTIONS:
Drug: MKC253 Inhalation Powder — Inhalation powder

SUMMARY:
26 subjects will be enrolled into 5 different dose groups. The trial will consist of a screening, a dosing and a follow-up visit.

Dosing at visit 2, of MKC253 Inhalation Powder, Glucagon-Like Peptide-1 (GLP-1) will be given at 5 dose levels.

DETAILED DESCRIPTION:
This Phase 1a , single-dose trial incorporates an open-label, ascending dose strategy to determine the safety & tolerability of MKC253 (GLP1/TechnosphereÂ®)Inhalation Powder.

The trial consists of a screening, dosing and a follow-up visit. Single dose administration of MKC253 occurs at the dosing visit. Five doses are being assessed: 0.05, 0.45, 0.75, 1.05 & 1.5 mg GLP-1. Dosing of each ascending cohort will occur after the Principal Investigator has reviewed all safety/tolerability data

ELIGIBILITY:
Inclusion Criteria:

* Healthy males = 18 and = 45 years of age
* Written Informed Consent.
* Body Mass Index (BMI) of < 30 kg/m2
* Non-smoker
* Normal pulmonary function and performance on pulmonary function tests

Exclusion Criteria:

* Clinically significant disease including diabetes mellitus
* Fasting blood glucose > 110 mg/dL (6.1 mmol/L)
* Significant psychiatric condition or drug or alcohol abuse
* Any other condition which, in the opinion of the PI, makes the subject unsuitable for the clinical trial, or could limit the validity of the informed consent and/or impair the subject's ability to participate in the trial
* Inability to perform PFT maneuvers meeting recommended American Thoracic Society (ATS) standards of acceptability and repeatability criteria

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2007-04; Primary Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Determine the safety and tolerability of ascending doses of MKC253 Inhalation Powder | 2 weeks

SECONDARY OUTCOMES:
Incidence of pulmonary and other AEs | 2 weeks
Pharmacokinetic (PK) parameters of plasma GLP-1 | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert Baughman, Study Director — Mannkind Corporation
Locations (1):
- University Medical Centre Groningen, Zuidlaren, Netherlands